CLINICAL TRIAL: NCT01580631
Title: Assessment of a Consensus Driven Narrow Band Imaging (NBI) Pattern Classification System in Barrett's Esophagus (BE)
Brief Title: Narrow Band Imaging Project on Barrett's Esophagus
Status: Suspended | Type: Observational
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, PRATEEK SHARMA, Principal Investigator, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Other Study IDs: PS0059
Record Dates: First submitted 2012-04-04; First posted 2012-04-19 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Barrett's Esophagus; Gastroesophageal Reflux Disease
Keywords: Narrow band imaging; Barrett's esophagus; Gastroesophageal reflux disease
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- BE with dysplasia.: Patients having Barrett's esophagus with dysplasia.
- BE without dysplasia.: Patients having Barrett's esophagus without dysplasia.

SUMMARY:
Narrow Band Imaging(NBI) improves image contrast by allowing the blue light centered at 415 nanometers which is heavily absorbed by oxyhemoglobin to highlight the tissue's microvasculature and enhances detail on the surface of the mucosa revealing subtle changes. Barrett's esophagus(BE) has the mucosal and vessel changes during cancer transformation by angiogenesis. The ability of the NBI scope to visualize submucosal vessels forms the premise for the prediction of dysplasia in BE mucosa.

NBI images of the BE mucosa obtained during endoscopy will be classified by academic endoscopists and community endoscopists initially. The endoscopists will then be asked to predict histopathology based on the NBI surface patterns. This clinical trial will evaluate the inter-observer agreement of a simple, consensus driven narrow band imaging (NBI) classification system of surface patterns and its ability to differentiate dysplastic versus non-dysplastic Barrett's esophagus(BE) in patients undergoing BE screening or surveillance in expert academic centers and in community GI practice as well. Their performance will be evaluated for accuracy, sensitivity, specificity, positive predictive value and negative predictive value of each pattern that is visualized on NBI.

DETAILED DESCRIPTION:
This is a multicenter, prospective, double-blinded study of NBI images from 50 patients enrolled in the study. Patients undergoing BE screening and BE surveillance will be enrolled into the study. After meeting eligibility criteria, and obtaining an informed consent, patients will undergo their routine upper endoscopic examination using white light endoscopy. During the course of the upper endoscopy, the BE surface patterns will be carefully examined with the endoscope in overview mode (with the endoscope in the center of the esophageal lumen) and then in close proximity to the BE surface (approximately 3-5 mm away from the mucosa). In each of these positions, a maximum of 4 high quality images will be obtained from different surface patterns initially with WLE and then using NBI. Image capture will be standardized. All the images will be classified based upon a simplified NBI classification system using two main criteria:(1)mucosal pattern(regular/irregular/uncertain) and (2)vascular pattern (regular/irregular/uncertain). All images will be captured using a high-definition, NBI endoscope (190 endoscopes-GIF-HQ 190 [dual focus],Olympus Inc) and stored in the high quality TIFF format. After images have been obtained, target biopsies will be obtained from each area and submitted for histopathological evaluation in separate jars. From the reports on NBI patterns from the images by Gastroenterologist and corresponding histopathological details, the accuracy and interobserver agreement of this NBI classification system will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients age: ≥ 18 years
* Undergoing endoscopy for surveillance or endoscopic treatment of Barrett's esophagus
* Ability to take oral proton pump inhibitor
* For female subjects of childbearing potential, a negative urine pregnancy test within 2 weeks of enrollment and any subsequent endoscopy encounter
* Subject is eligible for treatment and follow-up endoscopy and biopsy as required by the investigational plan
* Ability to discontinue Aspirin/NSAIDs/Clopidogrel 7 days before and after all ablation procedures
* Ability to provide written, informed consent and understands the responsibilities of trial participation

Exclusion Criteria:

* The subject is pregnant or planning a pregnancy during the study period (12 months after treatment)
* Esophageal stricture preventing passage of endoscope or catheter
* Active erosive esophagitis
* Prior endoscopic therapy with endoscopic mucosal resection, radiofrequency ablation, etc.
* History of esophageal varices or coagulopathy
* Prior radiation therapy to the esophagus, except head and neck region radiation therapy.
* Evidence of esophageal varices during treatment endoscopy
* Subject has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines
* The subject is currently enrolled in an investigational drug or device trial that clinically interferes with the current study.
* Subject suffers from psychiatric or other illness deemed by the investigator as an inability to comply with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects at the participating institution who meet the inclusion criteria for this study will be offered the opportunity to participate in this clinical trial.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-10; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Determine the inter-observer agreement of a consensus driven NBI classification system in Barrett's esophagus. | 12 months
  Identifying newer consensus driven NBI classification system in Barrett's esophagus for better inter observer agreement among experts and community/general gastroenterologists. Higher interobserver agreement (measured by Landis and Koch method) on these NBI patterns in Barrett's esophagus will help in diagnosing dysplasia in an uniform way among the gastroenterologists.

SECONDARY OUTCOMES:
Accuracy of the NBI patterns in predicting dysplasia in Barrett's esophagus based on confidence and image quality. | 12 months
  Accuracy of the newer patterns for diagnosing dysplasia in Barrett's esophagus based on confidence and image quality perceived by the reviewer.
Sensitivity of the newer NBI classification in identifying dysplasia in Barrett's esophagus. | 12 months
  Sensitivity of the newer NBI patterns in predicting dysplasia in Barrett's esophagus.
Specificity of the newer NBI classification in identifying dysplasia in Barrett's esophagus. | 12 months
  Specificity of the newer NBI patterns in predicting dysplasia in Barrett's esophagus.
Positive predictive value of the newer NBI classification in identifying dysplasia in Barrett's esophagus. | 12 months
  Positive predictive value of the newer NBI patterns in predicting dysplasia in Barrett's esophagus.
Negative predictive value of the newer NBI classification in identifying dysplasia in Barrett's esophagus. | 12 months
  Negative predictive value of the newer NBI patterns in predicting dysplasia in Barrett's esophagus.

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Kansas City VA Medical Center; Irving Waxman, MD, Principal Investigator — University of Chicago; Jacques Bergman, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc; Helmut Messman, MD, Principal Investigator — University of Regensburg; Kenichi Goda, MD, Principal Investigator — Jikei University; Motosugu Kato, MD, Principal Investigator — Hokkaido University
Locations (4):
- United States (2):
  - The University of Chicago Medical Center, Chicago, Illinois
  - Kansas City VA Medical Center, Kansas City, Missouri
- University of Regensburg, Augsburg, Germany
- Amsterdam Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Background] Reid BJ, Sanchez CA, Blount PL, Levine DS. Barrett's esophagus: cell cycle abnormalities in advancing stages of neoplastic progression. Gastroenterology. 1993 Jul;105(1):119-29. doi: 10.1016/0016-5085(93)90017-7. PMID 8514029
- [Background] Wang KK, Sampliner RE; Practice Parameters Committee of the American College of Gastroenterology. Updated guidelines 2008 for the diagnosis, surveillance and therapy of Barrett's esophagus. Am J Gastroenterol. 2008 Mar;103(3):788-97. doi: 10.1111/j.1572-0241.2008.01835.x. No abstract available. PMID 18341497
- [Background] Sharma P, McQuaid K, Dent J, Fennerty MB, Sampliner R, Spechler S, Cameron A, Corley D, Falk G, Goldblum J, Hunter J, Jankowski J, Lundell L, Reid B, Shaheen NJ, Sonnenberg A, Wang K, Weinstein W; AGA Chicago Workshop. A critical review of the diagnosis and management of Barrett's esophagus: the AGA Chicago Workshop. Gastroenterology. 2004 Jul;127(1):310-30. doi: 10.1053/j.gastro.2004.04.010. PMID 15236196
- [Background] Cooper GS, Kou TD, Chak A. Receipt of previous diagnoses and endoscopy and outcome from esophageal adenocarcinoma: a population-based study with temporal trends. Am J Gastroenterol. 2009 Jun;104(6):1356-62. doi: 10.1038/ajg.2009.159. Epub 2009 May 12. PMID 19491849
- [Background] Corley DA, Levin TR, Habel LA, Weiss NS, Buffler PA. Surveillance and survival in Barrett's adenocarcinomas: a population-based study. Gastroenterology. 2002 Mar;122(3):633-40. doi: 10.1053/gast.2002.31879. PMID 11874995
- [Background] Sharma P, Falk GW, Weston AP, Reker D, Johnston M, Sampliner RE. Dysplasia and cancer in a large multicenter cohort of patients with Barrett's esophagus. Clin Gastroenterol Hepatol. 2006 May;4(5):566-72. doi: 10.1016/j.cgh.2006.03.001. Epub 2006 Apr 17. PMID 16630761
- [Background] Inadomi JM, Sampliner R, Lagergren J, Lieberman D, Fendrick AM, Vakil N. Screening and surveillance for Barrett esophagus in high-risk groups: a cost-utility analysis. Ann Intern Med. 2003 Feb 4;138(3):176-86. doi: 10.7326/0003-4819-138-3-200302040-00009. PMID 12558356
- [Background] Inadomi JM. Surveillance in Barrett's esophagus: a failed premise. Keio J Med. 2009 Mar;58(1):12-8. doi: 10.2302/kjm.58.12. PMID 19398879
- [Background] Falk GW, Rice TW, Goldblum JR, Richter JE. Jumbo biopsy forceps protocol still misses unsuspected cancer in Barrett's esophagus with high-grade dysplasia. Gastrointest Endosc. 1999 Feb;49(2):170-6. doi: 10.1016/s0016-5107(99)70482-7. PMID 9925694
- [Background] Reid BJ, Blount PL, Feng Z, Levine DS. Optimizing endoscopic biopsy detection of early cancers in Barrett's high-grade dysplasia. Am J Gastroenterol. 2000 Nov;95(11):3089-96. doi: 10.1111/j.1572-0241.2000.03182.x. PMID 11095322
- [Background] Egger K, Werner M, Meining A, Ott R, Allescher HD, Hofler H, Classen M, Rosch T. Biopsy surveillance is still necessary in patients with Barrett's oesophagus despite new endoscopic imaging techniques. Gut. 2003 Jan;52(1):18-23. doi: 10.1136/gut.52.1.18. PMID 12477753